CLINICAL TRIAL: NCT00296777
Title: Medication Treatment Following Neuropsychologic, Dichotic and f-MRI Tests in Depressed Outpatients With Repeat f-MRI Following Treatment
Brief Title: Treatment of Depression Following Multiple Brain Tests
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: #4781
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Major Depression; Dysthymia
Keywords: Major Depression; Dysthymia; f-MRI; Escitalopram; Bupropion; Imipramine; Neuropsychologic test; Dichotic listening; EEG; ERP
MeSH Terms: conditions — Depressive Disorder, Major; Dysthymic Disorder | interventions — Escitalopram; Bupropion; Imipramine; dimethophrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- escitalopram (Experimental): escitalopram 10 mg/d, increasing by 10 mg/week if tolerated and not remitted to maximum dose of 40 mg/d
  Interventions: Drug: Escitalopram
- bupropion (Experimental): bupropion XL 150 mg/d, increasing by 150 mg/d if tolerated and not remitted to maximum dose of 450 mg/d
  Interventions: Drug: Bupropion
- imipramine (Experimental): imipramine 50 mg/d for 3 days, then 100 mg/d for 4 days, then 150 mg/d for 3 days then 200 mg/d for 4 days then 250 mg/d for a week and then 300 mg/d thereafter, all dose increases if tolerated and not remitted
  Interventions: Drug: Imipramine

INTERVENTIONS:
Drug: Escitalopram — 8 weeks: up to 40 mg/day
  Other Names: Lexapro
  Arms: escitalopram
Drug: Bupropion — 8 weeks: up to 450 mg/day (for patients without history of seizures or risk for developing seizures.
  Other Names: Wellbutrin
  Arms: bupropion
Drug: Imipramine — 8 weeks: up to 300mg/day
  *if patient does not have contraindication.
  Other Names: Tofranil, Pressamine
  Arms: imipramine

SUMMARY:
The main purpose of this study is to correlate brain testing with treatment outcome.

DETAILED DESCRIPTION:
40 medication-free Depressed Patients will receive a battery of neuropsychologic tests, standard dichotic listening tests, EEG, ERP and an f-MRI while performing a neuropsychologic test, the Simon. Once testing is completed, patients will be treated in an open treatment trial of SSRI. Non-responders will then receive Bupropion followed by Tricyclic Antidepressant if still depressed. While our main purpose is to correlate imaging testing with other measures of brain functioning, we also intend to see whether f-MRI findings demonstrate specific brain areas which differ between responders and non-responders. At the end of SSRI treatment, patients will have a second f-MRI scan to investigate any changes treatment and/or response may have caused.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV Major Depression or Dysthymia
* Age 18-65
* Physically healthy
* Normal hearing
* Drug-free (two weeks for most antidepressants, four weeks for Fluoxetine)

Exclusion Criteria:

* Hearing deficit in one or both ears
* Body metal (e.g., wire stitches, screws in bones, stainless steel hips)
* History of Psychosis or Epilepsy
* Current (past six months) Substance Use Disorder (illicit drugs and/or alcohol)
* Unstable medical problem
* Insufficient English for neuropsychological and dichotic testing
* Bipolar I
* Need for wash-out from effective treatment in order to participate
* Pregnant
* High suicide risk
* Currently taking (within 2 weeks; 4 weeks for Fluoxetine) antidepressants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-12; Primary Completion 2007-05 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Scale (HAM-D) | 7 mos.

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | 7 mos.
Clinical Global Impression (CGI) | 7 mos.
Patient Global Impression (PGI) | 7 mos.
Inventory of Depressive Symptoms (IDS) | 7 mos.
Edinburgh Handedness Inventory | 7 mos.
Chapman Pleasure Scale | 7 mos.
Spielberger State/Trait Anxiety Inventory | 7 mos.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W. Stewart, MD., Principal Investigator — New York State Psychiatric Institute - Columbia University Department of Psychiatry
Locations (1):
- Depression Evaluation Service - New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Background] Taylor BP, Bruder GE, Stewart JW, McGrath PJ, Halperin J, Ehrlichman H, Quitkin FM. Psychomotor slowing as a predictor of fluoxetine nonresponse in depressed outpatients. Am J Psychiatry. 2006 Jan;163(1):73-8. doi: 10.1176/appi.ajp.163.1.73. PMID 16390892
- [Background] Bruder GE, Stewart JW, Voglmaier MM, Harrison WM, McGrath P, Tricamo E, Quitkin FM. Cerebral laterality and depression: relations of perceptual asymmetry to outcome of treatment with tricyclic antidepressants. Neuropsychopharmacology. 1990 Feb;3(1):1-10. PMID 2306330
- [Background] Bruder GE, Otto MW, McGrath PJ, Stewart JW, Fava M, Rosenbaum JF, Quitkin FM. Dichotic listening before and after fluoxetine treatment for major depression: relations of laterality to therapeutic response. Neuropsychopharmacology. 1996 Aug;15(2):171-9. doi: 10.1016/0893-133X(95)00180-L. PMID 8840353
- [Background] Stewart JW, Quitkin FM, McGrath PJ, Bruder GE. Do tricyclic responders have different brain laterality? J Abnorm Psychol. 1999 Nov;108(4):707-10. doi: 10.1037//0021-843x.108.4.707. PMID 10609436
- [Background] Bruder GE, Stewart JW, Tenke CE, McGrath PJ, Leite P, Bhattacharya N, Quitkin FM. Electroencephalographic and perceptual asymmetry differences between responders and nonresponders to an SSRI antidepressant. Biol Psychiatry. 2001 Mar 1;49(5):416-25. doi: 10.1016/s0006-3223(00)01016-7. PMID 11274653
- [Background] Bruder GE, Stewart JW, McGrath PJ, Deliyannides D, Quitkin FM. Dichotic listening tests of functional brain asymmetry predict response to fluoxetine in depressed women and men. Neuropsychopharmacology. 2004 Sep;29(9):1752-61. doi: 10.1038/sj.npp.1300519. PMID 15238992
- See also: Depression Evaluation Service - official website — http://www.depression-nyc.org
- See also: New York State Psychiatric Institute - official website — http://www.nyspi.org